CLINICAL TRIAL: NCT05424822
Title: A Phase 1, First-in-human Study of JNJ-80948543, a T-cell Redirecting Antibody, in Participants With NHL and CLL
Brief Title: A Study of JNJ-80948543, a T-cell Redirecting CD79b x CD20 x CD3 Trispecific Antibody, in Participants With Non-Hodgkin Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR109174; 2022-000685-18 (EudraCT Number); 80948543LYM1001 (Other: Janssen Research & Development, LLC); 2023-504187-42-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation (Experimental): Participants will receive JNJ-80948543 either by subcutaneous (SC) or intravenous (IV) administration to determine the putative recommended Phase 2 dose (RP2D) dosing schedule(s) and route(s) of administration based on safety, pharmacokinetic, pharmacodynamic, and preliminary assessment of efficacy across several dose regimens.
  Interventions: Drug: JNJ-80948543
- Part B: Cohort Expansion (Experimental): Participants will receive JNJ-80948543 by SC or IV administration.
  Interventions: Drug: JNJ-80948543

INTERVENTIONS:
Drug: JNJ-80948543 — JNJ-80948543 will be administered as SC or IV injection.

SUMMARY:
The purpose of this study is to characterize safety and to determine the putative recommended Phase 2 dose(s) (RP2D[s]), optimal dosing schedule(s) and route(s) of administration of JNJ-80948543 in Part A (Dose Escalation) and to further characterize the safety of JNJ-80948543 at the putative RP2D(s) in Part B (Cohort Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of disease: B-cell non-Hodgkin lymphoma (NHL) or chronic lymphocytic leukemia (CLL) requiring therapy.

All participants must have relapsed or refractory disease with no other approved therapies available that would be more appropriate in the investigator's judgment.

B-cell NHL as defined per the 2016 world health organization (WHO) classification. In addition, the following disease-specific criteria outlined below must be met:

If diffuse large B-cell lymphoma (DLBCL) or other high-Grade B-cell lymphoma: Received, or not eligible for high-dose chemotherapy and autologous stem cell transplantation with curative intent or deemed not eligible or fit for an alternative 2nd line therapy. Participants may be eligible if relapsing after chimeric antigen receptors (CAR-T) cell treatment or while waiting for a CAR-T cell treatment.

If transformed lymphoma from low Grade B-cell malignancies: Received or not a candidate for an approved first-line regimen for DLBCL and received or not eligible for high-dose chemotherapy and autologous stem cell transplantation with curative intent.

If follicular lymphoma (FL) (all grades): Previously treated with a minimum of 2 prior lines of systemic therapy, with at least one prior line containing an anti-CD20 antibody.

If mantle cell lymphoma (MCL), marginal zone lymphoma (MZL) (including nodal, extranodal/MALT, and splenic MZL subtypes): Previously treated with at least 2 lines of systemic therapy. H.pylori-positive gastric MALT lymphoma must have failed prior H. pylori eradication therapy as one of their prior lines .

Waldenstrom macroglobulinemia (WM): Previously treated with at least 1 line of systemic therapy.

small lymphocytic lymphoma/chronic lymphocytic leukemia (CLL/SLL): Relapsed or refractory with at least 2 prior lines of therapy, including a Bruton tyrosine kinase inhibitor (BTK) inhibitor or a BCL2 inhibitor, if eligible. In addition for part B Participants must have measurable disease as defined by the appropriate disease response criteria

* Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0 or 1
* Cardiac parameters within the following range: corrected QT interval (QTc intervals corrected using Fridericia's formula [QTcF]) less than or equal to (<=) 480 milliseconds based on the average of triplicate assessments performed no more than 5 (plus minus [+-] 3) minutes apart
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (beta- human chorionic gonadotropin) at screening and must agree to further serum or urine pregnancy tests prior to the first dose, during the study and until 3 months after the last dose of study treatment
* A female participant must agree not to be pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 3 months after the last dose of study treatment

Exclusion Criteria:

* Known active central nervous system (CNS) involvement; Lymphoma with CNS involvement may be allowed in pharmacokinetic/ pharmacodynamic (PK/PD) and expansion cohorts if approved by the study evaluation team (SET)
* Prior solid-organ transplantation
* Autoimmune or inflammatory disease requiring systemic steroids or other immunosuppressive agents (example, methotrexate or tacrolimus) within 1 year prior to first dose of study drug
* Toxicity from prior anticancer therapy has not resolved to baseline levels or to Grade <= 1 (except alopecia, vitiligo, peripheral neuropathy, or endocrinopathies that are stable on hormone replacement, which may be Grade 2)
* Clinically significant pulmonary compromise, particularly the need for supplemental oxygen use to maintain adequate oxygenation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicity (DLT) | Up to 4 Years 3 months
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.
Number of Participants with Adverse Events (AEs) | Up to 4 Years 3 months
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants with AE by Severity | Up to 4 Years 3 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE). Severity scale ranges from Grade 1 (Mild) to Grade 4 (Life-threatening). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event. Cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) will be graded as per American Society for Transplantation and Cellular Therapy (ASTCT).

SECONDARY OUTCOMES:
Serum Concentration of JNJ-80948543 | Up to 4 Years 3 months
  Serum samples will be analyzed to determine concentrations of JNJ-80948543 using a validated, specific, and sensitive method.
Number of Participants with Presence of Anti-Drug Antibodies of JNJ-80948543 | Up to 4 Years 3 months
  Number of participants with presence of anti-drug antibodies of JNJ-80948543 will be assessed.
Overall Response Rate (ORR) | Up to 4 Years 3 months
  ORR is defined as the percentage of participants who have a best response of partial response (PR) or better.
Complete Response (CR) Rate | Up to 4 Years 3 months
  CR rate is defined as the percentage of participants who achieve a best response of CR.
Rate of VGPR or Better for Participants with Waldenstrom Macroglobulinemia (WM) | Up to 4 Years 3 months
  The response criteria planned to be used for participants with WM includes a category of VGPR, which is clinically understood to be better than PR but not as good as CR. For participants with WM, this rate is defined as the proportion of participants who achieve a best response of VGPR or better.
Time to Response (TTR) | Up to 4 Years 3 months
  TTR is defined for participants who achieved PR or CR as the time from the first dose of study drug to first response of PR or CR.
Duration of Response (DOR) | Up to 4 Years 3 months
  DOR is defined for participants who achieved a response of PR or better as the time between the date of initial documentation of first response of PR or better to the date of first documented evidence of progressive disease or death.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (29):
- United States (7):
  - City of Hope, Duarte, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (4):
  - Macquarie University Hospital, Macquarie University
  - The Alfred Hospital, Melbourne
  - Linear Clinical Research Ltd, Nedlands
  - Scientia Clinical Research, Randwick
- China (4):
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - Tianjin cancer hospital, Tianjin
  - Union Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- France (4):
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Institut Curie, Paris
  - Institut de Cancerologie Strasbourg Europe ICANS, Strasbourg
  - Institut Universitaire du cancer de Toulouse-Oncopole, Toulouse
- Israel (3):
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa
  - Aichi Cancer Center, Nagoya
  - The Cancer Institute Hospital of JFCR, Tokyo
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne Osrodek Badan Klinicznych Wczesnych Faz, Gdansk
  - Aidport Sp z o o, Skorzewo

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency